CLINICAL TRIAL: NCT03991273
Title: Testing the Implementation Efficacy of Movement-to-Music Delivered in a Community-Based Fitness Center and Blended Onsite and Home-based Group Teleexercise Class: A Mixed-Methods Pilot Study.
Brief Title: Testing the Implementation of Movement-to-Music in a Community Fitness Center and Blended Onsite and Teleexercise Class
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant projects were revised in response to COVID-19.
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Lakeshore Foundation (Other)
Responsible Party: Principal Investigator, Byron Lai, Project Coordinator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 90DPGE0005-01-00
Record Dates: First submitted 2019-06-13; First posted 2019-06-19 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Exercise; Disability Physical
Keywords: disability; disabilities; teleexercise; movement-to-music; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Y-M2M© (Experimental): a group-based M2M© program conducted onsite at a local YMCA
  Interventions: Other: Y-M2M©
- B-M2M© (Experimental): a blended program that provides Y-M2M© and a home-based M2M© via videoconferencing
  Interventions: Other: Y-M2M©; Other: B-M2M©

INTERVENTIONS:
Other: Y-M2M© — The Y-M2M© group will receive classes that will be delivered onsite at a YMCA facility. Movement-to-Music (M2M©) is an instructor-guided exercise program that is coupled with music to enhance strength, cardiorespiratory capacity, range of motion, and balance.
Other: B-M2M© — The B-M2M© group will receive the same onsite M2M© classes as the Y-M2M© group, but they will also be provided with the option of performing home-based M2M© that will be delivered via videoconferencing.
  Arms: B-M2M©

SUMMARY:
To prepare for a large scale-up study, the goal of this pilot implementation trial is to examine the feasibility of Movement-to-Music (M2M©) delivery mechanisms through two channels: 1) a group-based M2M© program conducted onsite at a local YMCA; and 2) a blended program that provides Y-M2M© and a home-based M2M© (B-M2M©) via videoconferencing. A key element of this pilot is to examine issues associated with participant-provider interactions, and to better understand the robustness of the technology to deliver a group-based (teleexercise) version of M2M© in the home setting.

DETAILED DESCRIPTION:
There will be 4 phases to this study. In phase 1, the investigators will explore potential barriers and supports that may affect the delivery of M2M© at one YMCA facility through one-on-one interviews with YMCA staff that have been trained to conduct M2M©.

Phase 2 will include a quantitative monitoring phase. During this phase the 2 delivery mechanisms of M2M© (Y-M2M© and B-M2M©) will be evaluated through assessments of quantitative feasibility metrics before, during, and after the intervention. The intervention will include a convenient sample of 54 participants.

To expand on the findings from the previous quantitative phase, phase 3 will include post-intervention focus group interviews conducted separately for each stakeholder group: all 54 participants, M2M© trainers, research assistants involved with technical support, and YMCA staff that were involved with the project.

During phase 4 (the integrative phase), the researchers will compile the quantitative and qualitative findings for the three primary feasibility metrics (process, resource, and management). These findings will then be comprehensively analyzed by a review panel that will provide suggestions for improvement within each metric. The panel will then discuss the summative findings and vote towards acceptable or not acceptable feasibility.

The 12-week Y-M2M© intervention will be pilot tested at one YMCA facility in Birmingham, AL.The B-M2M© group will be provided with the flexibility of attending the same onsite classes at the YMCA facility as participants in the Y-M2M© group and will also be able to participate in group M2M© teleexercise classes at home that are conducted through Internet video conferencing.

The investigators will use a permuted block randomization design to ensure close balance between the arms across waves and to increase the unpredictability in the upcoming assignment and prevent inadvertent bias. The project statistician will generate the randomization list that will be provided to the project coordinator in sealed envelopes to conceal the allocation. Assessors (health and function assessments done at Lakeshore Foundation) will be blinded to participant assignment and allocation of the arm assignment will not be done until baseline testing and measures are collected.

Primary quantitative outcomes will include those related to process, resources, and management. In summary, these metrics will include measures of adherence, issues that arise with implementation and the efficiency to which they are resolved, and intervention fidelity between the delivery sites. Secondary quantitative outcomes will include estimates of variability in scientific outcomes (physical activity; quality of life; social participation; fitness Measures (cardiorespiratory fitness, muscle strength, lower extremity function; social cognitive theory constructs [Self-efficacy, Outcome expectations, Barriers, Social support]).

ELIGIBILITY:
Inclusion Criteria:

1. primary diagnosis of head injury, stroke, MS, spinal cord injury, spina bifida, Parkinson's disease or cerebral palsy conferred by a physician and fits one of the three functional mobility groups (Groups I-III);
2. between the ages of 19 to 70 yrs.;
3. physician clearance to participate;
4. willing to participate in an exercise program 3 times per week;
5. conversant in and reads English.

Exclusion Criteria:

1. participated in a similar intervention in the last 6 months;
2. use of tobacco products in the last 6 months;
3. cognitive impairment;
4. active pressure ulcer;
5. any contraindications to exercise based on the American College of Sports Medicine (ACSM) guidelines;
6. visual acuity that prevents following a group exercise class;
7. significant hearing impairment impeding ability to hear music to engage in exercise.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-20 (Estimated); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Phase 1: Foreseeable implementation barriers and supports as reported by YMCA trainers | Pre-intervention (week 0)
  Prior to conducting the intervention, the investigators will conduct interviews to qualitatively explore YMCA trainers' perceptions of organizational or system factors that can potentially facilitate the adoption of M2M© in YMCAs and tailor the M2M© delivery plan accordingly (using open-ended questions).
Phase 2: Quantitative feasibility metric (Process outcome #1:Enrollment Rate) | Intervention (weeks 1-12)
  Enrollment rate: the number of participants screened / total enrolled
Phase 2: Quantitative feasibility metric (Process outcome #2: Class Attendance) | Intervention (weeks 1-12)
  Attendance to the exercise sessions: total number of sessions attended divided by the total 36 prescribed sessions
Phase 2: Quantitative feasibility metric (Process outcome #3: Attrition Rate) | Intervention (weeks 1-12)
  Attrition rate: number of participants that withdraw from the intervention
Phase 2: Quantitative feasibility metric (Process outcome #4: Time to complete data collection) | Intervention (weeks 1-12)
  Time to complete data collection: time in minutes required to complete data collection (average of both pre- and post-data collection visit times)
Phase 2: Quantitative feasibility metric (Process outcome #1: Technical difficulties with technology) | Intervention (weeks 1-12)
  Technical difficulties with technology: Frequency of issues experienced by participants and trainers
Phase 2: Quantitative feasibility metric (Resource outcome #2: Resources required by the YMCA) | Intervention (weeks 1-12)
  Resources required by the YMCA: # of items purchased for a YMCA M2M class
Phase 2: Quantitative feasibility metric (Management outcome #1: M2M fidelity between conditions) | Intervention (weeks 1-12)
  M2M fidelity between conditions: the frequency of times a deviation from the protocol was observed for both the YMCA and Teleexercise classes.
Phase 2: Quantitative feasibility metric (Management outcome #2: Issues with data management) | Intervention (weeks 1-12)
  Issues with data management: frequency of issues encountered
Phase 3: Qualitative interview exploring stakeholders' perceptions of intervention implementation | Post-Intervention (week 13)
  Focus group interviews will be conducted separately for each stakeholder group: all 54 participants, M2M© trainers, research assistants involved with technical support, and YMCA staff that were involved with the project. The semi-structured interviews will explore participants' perceptions regarding the intervention implementation process, resources, and management (using open-ended questions)

SECONDARY OUTCOMES:
Phase 2: Quantitative feasibility metric (Scientific outcome #1: Physical Activity) | Intervention (weeks 1 and 12)
  Physical Activity: measured via the Godin Leisure-Time Exercise Questionnaire (total score and health-contribution score)
Phase 2: Quantitative feasibility metric (Scientific outcome #2: Quality of life) | Intervention (weeks 1 and 12)
  Quality of life: measured via the NIH PROMIS 10 Global Health Items (total score)
Phase 2: Quantitative feasibility metric (Scientific outcome #3: Social participation) | Intervention (weeks 1 and 12)
  Social participation: measured via the NIH PROMIS Ability to Participate in Social Roles and Activities
Phase 2: Quantitative feasibility metric (Scientific outcome # 4: Self-Efficacy) | Intervention (weeks 1 and 12)
  Self-Efficacy: measured via the Exercise Self-Efficacy Scale (total score)
Phase 2: Quantitative feasibility metric (Scientific outcome # 5: Outcome expectations) | Intervention (weeks 1 and 12)
  Outcome expectations: measured via the Multidimensional Outcomes Expectations for Exercise Scale (total score)
Phase 2: Quantitative feasibility metric (Scientific outcome # 6: Barriers) | Intervention (weeks 1 and 12)
  Barriers to physical activity: measured via the Barriers in Physical Activity Questionnaire (total score)
Phase 2: Quantitative feasibility metric (Scientific outcome # 7: Social support) | Intervention (weeks 1 and 12)
  Social support: measured via the Social Provision Scale (total score)
Phase 2: Quantitative feasibility metric (Scientific outcome # 8: Cardiorespiratory fitness) | Intervention (weeks 1 and 12)
  Cardiorespiratory fitness: peak oxygen consumption (ml.kg-1.min-1)
Phase 2: Quantitative feasibility metric (Scientific outcome # 9: Hand-grip strength) | Intervention (weeks 1 and 12)
  Cardiorespiratory fitness: peak hand-grip strength (Newtons; both hands)
Phase 2: Quantitative feasibility metric (Scientific outcome # 10: Lower extremity function) | Intervention (weeks 1 and 12)
  Lower extremity function: measured via the Short Physical Performance Battery (total score)
Phase 2: Quantitative feasibility metric (Scientific outcome # 11: Lower extremity function) | Intervention (weeks 1 and 12)
  Lower extremity function: measured via the Timed Up and Go (total score)

CONTACTS AND LOCATIONS:
Overall Officials: James H Rimmer, PhD, Study Chair — University of Alabama at Birmingham; Hui-Ju Young, PhD, Study Director — University of Alabama at Birmingham; Byron W Lai, PhD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: Yes
We will make a de-identified copy of the final data set available after we have completed the final analysis. We will make the data set available to the scientific community through the Inter-University Consortium for Political and Social Research account (which enables free downloads via Internet).
Supporting Information: Study Protocol
Time Frame: The data will be uploaded within 12 months of completing the study.
Access Criteria: Free downloads via the Internet
URL: https://www.icpsr.umich.edu/icpsrweb/